CLINICAL TRIAL: NCT04321967
Title: Topical Nitroglycerin as a Mechanism for Cutaneous Vaso-modulation and Improved Wound Healing After Breast Reduction
Brief Title: Nitropaste in Breast Reduction
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Unable to recruit patients
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Peter J. Taub, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCO 19-0387
Record Dates: First submitted 2020-03-24; First posted 2020-03-26 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2021-01

CONDITIONS: Gynecomastia; Delayed Wound Healing
Keywords: Nitroglycerin paste; Scarring; Necrosis; Wound healing; Breast; Breast reduction
MeSH Terms: conditions — Gynecomastia; Cicatrix; Necrosis | interventions — octyl 2-cyanoacrylate

STUDY DESIGN:
Intervention Model Description: Patients who agree to participate will be randomized during their bilateral breast reduction procedure. Each patient will be randomized to "LEFT BREAST" or "RIGHT BREAST." The randomization result will determine which breast receives the nitroglycerin paste. Their breast reduction will be done using the Wise pattern, and all incisions will be sealed with Dermabond. At the conclusion of the procedure, 1g of topical nitroglycerin (2%) will be placed on the breast which the randomizer indicated. Patients will be monitored for AEs during the remainder of their hospital stay.
Who Masked: Participant, Care Provider
Masking Description: The patient will be masked and will not know which breast received the nitropaste. The investigator who applied nitropaste will know which breast was treated, but the investigator who conducts the follow-up visits will not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nitroglycerine paste (Experimental): The randomized breast will receive Nitroglycerine paste and Dermabond.
  Interventions: Drug: Nitroglycerin Paste; Drug: Dermabond
- Dermabond (Placebo Comparator): The control breast will receive Dermabond only
  Interventions: Drug: Dermabond

INTERVENTIONS:
Drug: Nitroglycerin Paste — 1g of 2% Nitroglycerin paste topical application
  Arms: Nitroglycerine paste
Drug: Dermabond — Topical skin adhesive

SUMMARY:
The purpose of this study is evaluate the effect of Nitroglycerin paste on wound healing and scarring. Previous research has shown that Nitroglycerin paste can improve the blood flow to a wound, which may be associated with better wound healing, and ultimately, better scarring.

DETAILED DESCRIPTION:
This will be a single-center, patient-blinded, (breast) randomized trial utilizing nitroglycerin paste on their breast reduction scar. The study team aims to randomize 100 patients, or 200 breasts. Each patient will receive treatment, but the breast that received treatment will be random. This will allow for a control breast to compare to. Patients will be followed for 12 months postoperatively to observe wound healing.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are female and transmen
* Undergoing bilateral breast reduction via Mount Sinai Plastic Surgery Clinic
* Reduction must be performed via Wise incisional pattern

Exclusion Criteria:

* Patients who are male or transwomen
* Patients who are under 18 years of age

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Change in Vancouver Scar Scoring (VSS) | First post-op visit (0 weeks post op) and last visit at 12 months
  Change in Vancouver Scar Scoring at 12 as compared to first post visit. VSS is a standardized scar appearance protocol - full score from 0-13, with higher score indicating poorer health outcomes.

SECONDARY OUTCOMES:
Number of occurrences of wound breakdown | 12 months
  Change in number of occurrence of necrosis and/or wound breakdown at 12 months as compared to the first post-op visit
Number of side-effects of Nitroglycerin use | 12 months
  Side effects of nitroglycerine use measured as a composite of side effects which includes pre-syncope, syncope, chest pains and headache.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Taub, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD and related data dictionaries available. The PI does not plan to share data at the conclusion of the study beyond what is published